CLINICAL TRIAL: NCT05142267
Title: Stress and Opioid Misuse Risk: The Role of Endogenous Opioid and Endocannabinoid Mechanisms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Stephen Bruehl, PhD, Professor of Anesthesiology, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 210399; R01DA050334 (NIH)
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use Disorder; Back Pain; Stress
MeSH Terms: conditions — Opioid-Related Disorders; Back Pain | interventions — Oxycodone; Naloxone

STUDY DESIGN:
Intervention Model Description: The study will be a mixed between/within-subjects design with double-blind counterbalanced placebo-controlled administration of both an opioid antagonist and an opioid agonist. Both drugs are being administered solely to probe mechanisms linking stress with individual differences in opioid analgesic responses (this is not an efficacy trial).
Masking Description: The participant and investigator will be blinded to the drug order across the 3 laboratory drug administration sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adults with chronic non-cancer low back pain (Other)
  Interventions: Drug: Placebo; Drug: Oxycodone; Drug: Naloxone

INTERVENTIONS:
Drug: Placebo — In randomized order (crossover) across 3 laboratory sessions, participants will undergo laboratory evoked thermal pain response testing with: 1) 0.13 mg/kg of oral oxycodone (in 1mg/ml syrup) plus 20ml i.v. saline placebo, 2) 8mg of i.v. naloxone (in 20ml saline vehicle) plus oral placebo syrup (quantity matching oxycodone syrup volume), or 3) 20ml i.v. saline placebo plus oral placebo syrup (quantity matching oxycodone syrup volume).
  Thermal pain testing utilizes a Medoc TSAII NeuroSensory Analyzer. This equipment is used to assess heat pain threshold and tolerance using an ascending method of limits protocol.
  Other Names: normal saline placebo
Drug: Oxycodone — In randomized order (crossover) across 3 laboratory sessions, participants will undergo laboratory evoked thermal pain response testing with: 1) 0.13 mg/kg of oral oxycodone (in 1mg/ml syrup) plus 20ml i.v. saline placebo, 2) 8mg of i.v. naloxone (in 20ml saline vehicle) plus oral placebo syrup (quantity matching oxycodone syrup volume), or 3) 20ml i.v. saline placebo plus oral placebo syrup (quantity matching oxycodone syrup volume).
  Thermal pain testing utilizes a Medoc TSAII NeuroSensory Analyzer. This equipment is used to assess heat pain threshold and tolerance using an ascending method of limits protocol.
Drug: Naloxone — In randomized order (crossover) across 3 laboratory sessions, participants will undergo laboratory evoked thermal pain response testing with: 1) 0.13 mg/kg of oral oxycodone (in 1mg/ml syrup) plus 20ml i.v. saline placebo, 2) 8mg of i.v. naloxone (in 20ml saline vehicle) plus oral placebo syrup (quantity matching oxycodone syrup volume), or 3) 20ml i.v. saline placebo plus oral placebo syrup (quantity matching oxycodone syrup volume).
  Thermal pain testing utilizes a Medoc TSAII NeuroSensory Analyzer. This equipment is used to assess heat pain threshold and tolerance using an ascending method of limits protocol.
  Other Names: narcan

SUMMARY:
The purpose of this study is to see how stress influences the effects of opioid pain medications often used to help relieve back pain. The study will help to learn more about how high stress levels could increase risk for pain medication misuse.

DETAILED DESCRIPTION:
The purpose of this project is to advance mechanistic knowledge of how stress impacts differential opioid analgesic responses that enhance risk for opioid use disorder (OUD), potentially informing development of data-driven precision pain medicine algorithms to mitigate opioid related risks.

The study aims to determine whether subjective and physiological stress-related measures are associated with analgesic and misuse-relevant subjective responses to placebo-controlled oxycodone administration. The study also aims to evaluate associations between stress-related measures and both endogenous opioid (EO) function and endocannabinoid (EC) levels and to test whether EO and EC mechanisms contribute to associations between stress-related measures and oxycodone responses

Using a mixed between/within-subject design, the study will obtain baseline assessment of stress related markers followed by 3 laboratory sessions with assessment of endocannabinoids, back pain assessment, and exposure to standardized evoked pain stimuli after administration of placebo, naloxone, and oxycodone.

ELIGIBILITY:
Inclusion Criteria:

* Intact cognitive status and ability to provide informed consent
* Ability to read and write in English sufficiently to understand and complete study questionnaires (which are only validated in English)
* Age 18 or older And
* Presence of persistent daily low back pain of at least three months duration and of at least a 3/10 in average intensity

Exclusion Criteria:

* History of renal or hepatic dysfunction
* Reports of current or past alcohol or substance abuse or treatment for such condition
* A reported history of PTSD, psychotic, or bipolar disorders
* Chronic pain due to malignancy (e.g., cancer) or autoimmune disorders (e.g., rheumatoid arthritis, lupus)
* Reports of recent benzodiazepine use (confirmed via rapid urine screening prior to each lab session)
* Any medical conditions (e.g., significant cardiovascular disease) that the study physician feels would contraindicate participation in the lab stressors
* Reported daily opiate use within the past 6 months, or use of any opioid analgesic medications within 3 days of study participation (confirmed through rapid urine screening prior to each lab session)
* Pregnancy (females only, to avoid fetal drug exposure - pregnancy tests conducted prior to each lab session to confirm eligibility)
* Prior allergic reaction/intolerance to oxycodone or its analogs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Mean change in McGill Pain Questionnaire-2 (MPQ-2) ratings of low back pain from the placebo to oxycodone condition | Across 2 laboratory assessment days (an expected average of 15 day period)
  Mean within participant changes in McGill Pain Questionnaire-2 (MPQ-2) ratings of low back pain from the placebo to oxycodone condition (across 2 testing days). The MPQ-2 score ranges from 0-10 where 0 represents no pain and 10 represents most intense pain. Positive change values indicate decreased pain responsiveness post intervention.
Mean DELTA Drug Liking subscale scores in the oxycodone condition | One 1 laboratory assessment day
  Mean DELTA Drug Liking subscale scores in the oxycodone condition. The DELTA Drug Liking subscale consists of a single item asking about overall perceived drug liking. The 1-5 scale is anchored with 1 representing dislike a lot and 5 representing like a lot.
Composite measure of changes in MPQ-2 ratings of low back pain from the placebo to naloxone condition (standardized) plus plasma levels of endocannabinoids (standardized) | Across 2 laboratory assessment days (an expected average of 15 day period)
  Composite measure of changes in MPQ-2 ratings of low back pain from the placebo to naloxone condition (standardized) plus plasma levels of endocannabinoids (standardized). More negative standardized values will indicate low levels of endogenous pain inhibition and more positive levels will indicate high levels of endogenous pain inhibition.

SECONDARY OUTCOMES:
Mean changes in MPQ-2 ratings of ischemic task pain from the placebo to oxycodone condition | Across 2 laboratory assessment days (an expected average of 15 day period)
  Mean within participant changes in MPQ-2 ratings of ischemic task pain from the placebo to oxycodone condition. The MPQ-2 score ranges from 0-10 where 0 represents no pain and 10 represents most intense pain. Positive change values indicate decreased pain responsiveness.
Mean changes in Visual Analog Scale (VAS) intensity ratings of ischemic task pain from the placebo to oxycodone condition | Across 2 laboratory assessment days (an expected average of 15 day period)
  Mean within participant changes in VAS intensity ratings of ischemic task pain from the placebo to oxycodone condition. The score is a rating of current acute pain using a 0-100 visual analog scale (VAS) (0 = "no pain" and 100 = "worst possible pain")
Mean changes in MPQ-2 ratings of heat task pain from the placebo to oxycodone condition | Across 2 laboratory assessment days (an expected average of 15 day period)
  Mean within participant changes in MPQ-2 ratings of heat task pain from the placebo to oxycodone condition. The MPQ-2 score ranges from 0-10 where 0 represents no pain and 10 represents most intense pain. Positive change values indicate decreased pain responsiveness.
Mean changes in VAS intensity ratings of heat task pain from the placebo to oxycodone condition | Across 2 laboratory assessment days (an expected average of 15 day period)
  Mean within participant changes in VAS intensity ratings of heat task pain from the placebo to oxycodone condition. The score is a rating of current acute pain using a 0-100 visual analog scale (VAS) (0 = "no pain" and 100 = "worst possible pain")
DELTA Take Again subscale scores in the oxycodone condition | 1 laboratory assessment day (an expected average of 15 day period)
  Mean oxycodone condition Take Again (DELTA subscale) score. The score ranges from 1-5 where 1 represents definitely would not and 5 represents definitely would. Positive values indicate decreased overall drug effects post intervention.
Mean Delta Effects subscale in the oxycodone condition | 1 laboratory assessment day (an expected average of 15 day period)
  Mean oxycodone condition Effects (DELTA) -Drug Effect subscale ratings. The score ranges from 1-5 where 1 represents no effect and 5 represents very strong effect. Positive values indicate decreased overall drug effects post intervention.
Mean VAS Opioid Euphoria subscale in the oxycodone condition | 1 laboratory assessment day (an expected average of 15 day period)
  Mean oxycodone condition VAS Opioid Effects-Euphoria subscale ratings. The score ranges from 0-300 where 0 means no euphoria and 300 means most euphoria possible. Positive values indicate greater euphoria.
Mean VAS Opioid Unpleasantness subscale in the oxycodone condition | 1 laboratory assessment day (an expected average of 15 day period)
  Mean oxycodone condition VAS Opioid Effects-Unpleasantness subscale ratings. The score ranges from 0-300 where 0 means no unpleasantness and 300 means the most unpleasantness possible. Positive values indicate greater perceived unpleasantness.
Mean VAS Opioid Sedation subscale in the oxycodone condition | 1 laboratory assessment day (an expected average of 15 day period)
  Mean oxycodone condition VAS Opioid Effects-Sedation subscale ratings. The score ranges from 0-300 where 0 means no sedation and 300 means the most sedation possible. Positive values indicate greater sedation.
Mean change in McGill Pain Questionnaire-2 (MPQ-2) ratings of low back pain from the placebo to naloxone condition | Across 2 laboratory assessment days (an expected average of 15 day period)
  Mean within participant changes in McGill Pain Questionnaire-2 (MPQ-2) ratings of low back pain from the placebo to naloxone condition. The MPQ-2 score ranges from 0-10 where 0 represents no pain and 10 represents the most intense pain. Positive change values indicate greater endogenous opioid pain inhibition .
Mean change in McGill Pain Questionnaire-2 (MPQ-2) ratings of ischemic task pain from the placebo to naloxone condition | Across 2 laboratory assessment days (an expected average of 15 day period)
  Mean within participant changes in McGill Pain Questionnaire-2 (MPQ-2) ratings of ischemic task pain from the placebo to naloxone condition. The MPQ-2 score ranges from 0-10 where 0 represents no pain and 10 represents the most intense pain. Positive change values indicate greater endogenous opioid pain inhibition.
Mean changes in VAS intensity ratings of ischemic task pain from the placebo to naloxone condition | Across 2 laboratory assessment days (an expected average of 15 day period)
  Mean within participant changes in VAS intensity ratings of ischemic task pain from the placebo to naloxone condition. The VAS score is a rating of ischemic task pain using a 0-100 visual analog scale (VAS) (0 = "no pain" and 100 = "worst possible pain"). Positive change values indicate greater endogenous opioid pain inhibition.
Mean change in McGill Pain Questionnaire-2 (MPQ-2) ratings of heat task pain from the placebo to naloxone condition | Across 2 laboratory assessment days (an expected average of 15 day period)
  Mean within participant changes in McGill Pain Questionnaire-2 (MPQ-2) ratings of heat task pain from the placebo to naloxone condition. The MPQ-2 score ranges from 0-10 where 0 represents no pain and 10 represents the most intense pain. Positive change values indicate greater endogenous opioid pain inhibition
Mean changes in VAS intensity ratings of heat task pain from the placebo to naloxone condition | Across 2 laboratory assessment days (an expected average of 15 day period)
  Mean within participant changes in VAS intensity ratings of thermal task pain from the placebo to naloxone condition. The VAS score is a rating of ischemic task pain using a 0-100 visual analog scale (VAS) (0 = "no pain" and 100 = "worst possible pain"). Positive change values indicate greater endogenous opioid pain inhibition.
Mean plasma levels of endocannabinoids | Across 3 laboratory assessment days (an expected average of 15 day period)
  Mean plasma levels of endocannabinoids

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bruehl, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] al'Absi M, France C, Harju A, France J, Wittmers L. Adrenocortical and nociceptive responses to opioid blockade in hypertension-prone men and women. Psychosom Med. 2006 Mar-Apr;68(2):292-8. doi: 10.1097/01.psy.0000203240.64965.bd. PMID 16554396
- [Background] Altun A, Ozdemir E, Yildirim K, Gursoy S, Durmus N, Bagcivan I. The effects of endocannabinoid receptor agonist anandamide and antagonist rimonabant on opioid analgesia and tolerance in rats. Gen Physiol Biophys. 2015 Oct;34(4):433-40. doi: 10.4149/gpb_2015017. PMID 26374993
- [Background] Altun A, Yildirim K, Ozdemir E, Bagcivan I, Gursoy S, Durmus N. Attenuation of morphine antinociceptive tolerance by cannabinoid CB1 and CB2 receptor antagonists. J Physiol Sci. 2015 Sep;65(5):407-15. doi: 10.1007/s12576-015-0379-2. Epub 2015 Apr 18. PMID 25894754
- [Background] Baker TB, Piper ME, McCarthy DE, Majeskie MR, Fiore MC. Addiction motivation reformulated: an affective processing model of negative reinforcement. Psychol Rev. 2004 Jan;111(1):33-51. doi: 10.1037/0033-295X.111.1.33. PMID 14756584
- [Background] Bedse G, Hartley ND, Neale E, Gaulden AD, Patrick TA, Kingsley PJ, Uddin MJ, Plath N, Marnett LJ, Patel S. Functional Redundancy Between Canonical Endocannabinoid Signaling Systems in the Modulation of Anxiety. Biol Psychiatry. 2017 Oct 1;82(7):488-499. doi: 10.1016/j.biopsych.2017.03.002. Epub 2017 Mar 15. PMID 28438413
- [Background] Bluett RJ, Baldi R, Haymer A, Gaulden AD, Hartley ND, Parrish WP, Baechle J, Marcus DJ, Mardam-Bey R, Shonesy BC, Uddin MJ, Marnett LJ, Mackie K, Colbran RJ, Winder DG, Patel S. Endocannabinoid signalling modulates susceptibility to traumatic stress exposure. Nat Commun. 2017 Mar 28;8:14782. doi: 10.1038/ncomms14782. PMID 28348378
- [Background] Brat GA, Agniel D, Beam A, Yorkgitis B, Bicket M, Homer M, Fox KP, Knecht DB, McMahill-Walraven CN, Palmer N, Kohane I. Postsurgical prescriptions for opioid naive patients and association with overdose and misuse: retrospective cohort study. BMJ. 2018 Jan 17;360:j5790. doi: 10.1136/bmj.j5790. PMID 29343479
- [Background] Bruehl S, Burns JW, Chung OY, Quartana P. Anger management style and emotional reactivity to noxious stimuli among chronic pain patients and healthy controls: the role of endogenous opioids. Health Psychol. 2008 Mar;27(2):204-14. doi: 10.1037/0278-6133.27.2.204. PMID 18377139
- [Background] Bruehl S, Burns JW, Gupta R, Buvanendran A, Chont M, Kinner E, Schuster E, Passik S, France CR. Endogenous opioid function mediates the association between laboratory-evoked pain sensitivity and morphine analgesic responses. Pain. 2013 Sep;154(9):1856-1864. doi: 10.1016/j.pain.2013.06.002. Epub 2013 Jun 6. PMID 23748117
- [Background] Bruehl S, Burns JW, Gupta R, Buvanendran A, Chont M, Schuster E, France CR. Endogenous opioid inhibition of chronic low-back pain influences degree of back pain relief after morphine administration. Reg Anesth Pain Med. 2014 Mar-Apr;39(2):120-5. doi: 10.1097/AAP.0000000000000058. PMID 24553304
- [Background] Bruehl S, Burns JW, Morgan A, Koltyn K, Gupta R, Buvanendran A, Edwards D, Chont M, Kingsley PJ, Marnett L, Stone A, Patel S. The association between endogenous opioid function and morphine responsiveness: a moderating role for endocannabinoids. Pain. 2019 Mar;160(3):676-687. doi: 10.1097/j.pain.0000000000001447. PMID 30562268
- [Background] Bruehl S, Burns JW, Passik SD, Gupta R, Buvanendran A, Chont M, Schuster E, Orlowska D, France CR. The Contribution of Differential Opioid Responsiveness to Identification of Opioid Risk in Chronic Pain Patients. J Pain. 2015 Jul;16(7):666-75. doi: 10.1016/j.jpain.2015.04.001. Epub 2015 Apr 16. PMID 25892658
- [Background] Burns JW, Bruehl S, France CR, Schuster E, Orlowska D, Buvanendran A, Chont M, Gupta RK. Psychosocial factors predict opioid analgesia through endogenous opioid function. Pain. 2017 Mar;158(3):391-399. doi: 10.1097/j.pain.0000000000000768. PMID 27898491
- [Background] Carpenter RW, Lane SP, Bruehl S, Trull TJ. Concurrent and lagged associations of prescription opioid use with pain and negative affect in the daily lives of chronic pain patients. J Consult Clin Psychol. 2019 Oct;87(10):872-886. doi: 10.1037/ccp0000402. PMID 31556664
- [Background] Comer SD, Sullivan MA, Vosburg SK, Kowalczyk WJ, Houser J. Abuse liability of oxycodone as a function of pain and drug use history. Drug Alcohol Depend. 2010 Jun 1;109(1-3):130-8. doi: 10.1016/j.drugalcdep.2009.12.018. Epub 2010 Jan 15. PMID 20079977
- [Background] Crombie KM, Brellenthin AG, Hillard CJ, Koltyn KF. Endocannabinoid and Opioid System Interactions in Exercise-Induced Hypoalgesia. Pain Med. 2018 Jan 1;19(1):118-123. doi: 10.1093/pm/pnx058. PMID 28387833
- [Background] Dunne EM, Striley CW, Mannes ZL, Asken BM, Ennis N, Cottler LB. Reasons for Prescription Opioid Use While Playing in the National Football League as Risk Factors for Current Use and Misuse Among Former Players. Clin J Sport Med. 2020 Nov;30(6):544-549. doi: 10.1097/JSM.0000000000000628. PMID 29933284
- [Background] Griffiths RR, Bigelow GE, Ator NA. Principles of initial experimental drug abuse liability assessment in humans. Drug Alcohol Depend. 2003 Jun 5;70(3 Suppl):S41-54. doi: 10.1016/s0376-8716(03)00098-x. PMID 12759196
- [Background] Haller VL, Stevens DL, Welch SP. Modulation of opioids via protection of anandamide degradation by fatty acid amide hydrolase. Eur J Pharmacol. 2008 Dec 14;600(1-3):50-8. doi: 10.1016/j.ejphar.2008.08.005. Epub 2008 Aug 20. PMID 18762181
- [Background] Hassan AN, Le Foll B, Imtiaz S, Rehm J. The effect of post-traumatic stress disorder on the risk of developing prescription opioid use disorder: Results from the National Epidemiologic Survey on Alcohol and Related Conditions III. Drug Alcohol Depend. 2017 Oct 1;179:260-266. doi: 10.1016/j.drugalcdep.2017.07.012. Epub 2017 Aug 8. PMID 28818717
- [Background] Kavushansky A, Kritman M, Maroun M, Klein E, Richter-Levin G, Hui KS, Ben-Shachar D. beta-endorphin degradation and the individual reactivity to traumatic stress. Eur Neuropsychopharmacol. 2013 Dec;23(12):1779-88. doi: 10.1016/j.euroneuro.2012.12.003. Epub 2013 Jan 23. PMID 23352317
- [Background] Koob GF, Le Moal M. Addiction and the brain antireward system. Annu Rev Psychol. 2008;59:29-53. doi: 10.1146/annurev.psych.59.103006.093548. PMID 18154498
- [Background] Koob GF, Volkow ND. Neurobiology of addiction: a neurocircuitry analysis. Lancet Psychiatry. 2016 Aug;3(8):760-773. doi: 10.1016/S2215-0366(16)00104-8. PMID 27475769
- [Background] Lovallo WR, Acheson A, Vincent AS, Sorocco KH, Cohoon AJ. Early life adversity diminishes the cortisol response to opioid blockade in women: Studies from the Family Health Patterns project. PLoS One. 2018 Oct 12;13(10):e0205723. doi: 10.1371/journal.pone.0205723. eCollection 2018. PMID 30312327
- [Background] Lovallo WR, Enoch MA, Acheson A, Cohoon AJ, Sorocco KH, Hodgkinson CA, Vincent AS, Glahn DC, Goldman D. Cortisol Stress Response in Men and Women Modulated Differentially by the Mu-Opioid Receptor Gene Polymorphism OPRM1 A118G. Neuropsychopharmacology. 2015 Oct;40(11):2546-54. doi: 10.1038/npp.2015.101. Epub 2015 Apr 16. PMID 25881118
- [Background] Mayo LM, Asratian A, Linde J, Holm L, Natt D, Augier G, Stensson N, Vecchiarelli HA, Balsevich G, Aukema RJ, Ghafouri B, Spagnolo PA, Lee FS, Hill MN, Heilig M. Protective effects of elevated anandamide on stress and fear-related behaviors: translational evidence from humans and mice. Mol Psychiatry. 2020 May;25(5):993-1005. doi: 10.1038/s41380-018-0215-1. Epub 2018 Aug 17. PMID 30120421
- [Background] McCubbin JA, Bruehl S, Wilson JF, Sherman JJ, Norton JA, Colclough G. Endogenous opioids inhibit ambulatory blood pressure during naturally occurring stress. Psychosom Med. 1998 Mar-Apr;60(2):227-31. doi: 10.1097/00006842-199803000-00020. PMID 9560874
- [Background] McCubbin JA, Cheung R, Montgomery TB, Bulbulian R, Wilson JF. Aerobic fitness and opioidergic inhibition of cardiovascular stress reactivity. Psychophysiology. 1992 Nov;29(6):687-97. doi: 10.1111/j.1469-8986.1992.tb02047.x. PMID 1334271
- [Background] McCubbin JA, Surwit RS, Williams RB Jr. Endogenous opiate peptides, stress reactivity, and risk for hypertension. Hypertension. 1985 Sep-Oct;7(5):808-11. doi: 10.1161/01.hyp.7.5.808. PMID 4030048
- [Background] McCubbin JA, Wilson JF, Bruehl S, Ibarra P, Carlson CR, Norton JA, Colclough GW. Relaxation training and opioid inhibition of blood pressure response to stress. J Consult Clin Psychol. 1996 Jun;64(3):593-601. doi: 10.1037//0022-006x.64.3.593. PMID 8698954
- [Background] Morena M, Patel S, Bains JS, Hill MN. Neurobiological Interactions Between Stress and the Endocannabinoid System. Neuropsychopharmacology. 2016 Jan;41(1):80-102. doi: 10.1038/npp.2015.166. Epub 2015 Jun 12. PMID 26068727
- [Background] da Fonseca Pacheco D, Klein A, de Castro Perez A, da Fonseca Pacheco CM, de Francischi JN, Duarte ID. The mu-opioid receptor agonist morphine, but not agonists at delta- or kappa-opioid receptors, induces peripheral antinociception mediated by cannabinoid receptors. Br J Pharmacol. 2008 Jul;154(5):1143-9. doi: 10.1038/bjp.2008.175. Epub 2008 May 12. PMID 18469844
- [Background] Pacheco Dda F, Klein A, Perez AC, Pacheco CM, de Francischi JN, Reis GM, Duarte ID. Central antinociception induced by mu-opioid receptor agonist morphine, but not delta- or kappa-, is mediated by cannabinoid CB1 receptor. Br J Pharmacol. 2009 Sep;158(1):225-31. doi: 10.1111/j.1476-5381.2009.00310.x. Epub 2009 Jul 7. PMID 19594755
- [Background] Rougemont-Bucking A, Grazioli VS, Marmet S, Daeppen JB, Lemoine M, Gmel G, Studer J. Non-medical use of prescription drugs by young men: impact of potentially traumatic events and of social-environmental stressors. Eur J Psychotraumatol. 2018 May 9;9(1):1468706. doi: 10.1080/20008198.2018.1468706. eCollection 2018. PMID 29760868
- [Background] Sagar DR, Gaw AG, Okine BN, Woodhams SG, Wong A, Kendall DA, Chapman V. Dynamic regulation of the endocannabinoid system: implications for analgesia. Mol Pain. 2009 Oct 8;5:59. doi: 10.1186/1744-8069-5-59. PMID 19814807
- [Background] Salio C, Fischer J, Franzoni MF, Mackie K, Kaneko T, Conrath M. CB1-cannabinoid and mu-opioid receptor co-localization on postsynaptic target in the rat dorsal horn. Neuroreport. 2001 Dec 4;12(17):3689-92. doi: 10.1097/00001756-200112040-00017. PMID 11726775
- [Background] Shonesy BC, Bluett RJ, Ramikie TS, Baldi R, Hermanson DJ, Kingsley PJ, Marnett LJ, Winder DG, Colbran RJ, Patel S. Genetic disruption of 2-arachidonoylglycerol synthesis reveals a key role for endocannabinoid signaling in anxiety modulation. Cell Rep. 2014 Dec 11;9(5):1644-1653. doi: 10.1016/j.celrep.2014.11.001. Epub 2014 Nov 26. PMID 25466252
- [Background] Walsh SL, Nuzzo PA, Lofwall MR, Holtman JR Jr. The relative abuse liability of oral oxycodone, hydrocodone and hydromorphone assessed in prescription opioid abusers. Drug Alcohol Depend. 2008 Dec 1;98(3):191-202. doi: 10.1016/j.drugalcdep.2008.05.007. Epub 2008 Jul 7. PMID 18606504
- [Background] Welch SP. Interaction of the cannabinoid and opioid systems in the modulation of nociception. Int Rev Psychiatry. 2009 Apr;21(2):143-51. doi: 10.1080/09540260902782794. PMID 19367508
- [Background] Welch SP, Eads M. Synergistic interactions of endogenous opioids and cannabinoid systems. Brain Res. 1999 Nov 27;848(1-2):183-90. doi: 10.1016/s0006-8993(99)01908-3. PMID 10612710
- [Background] Wightman R, Perrone J, Portelli I, Nelson L. Likeability and abuse liability of commonly prescribed opioids. J Med Toxicol. 2012 Dec;8(4):335-40. doi: 10.1007/s13181-012-0263-x. PMID 22992943
- [Background] Younger JW, Lawler-Row KA, Moe KA, Kratz AL, Keenum AJ. Effects of naltrexone on repressive coping and disclosure of emotional material: a test of the opioid-peptide hypothesis of repression and hypertension. Psychosom Med. 2006 Sep-Oct;68(5):734-41. doi: 10.1097/01.psy.0000234029.38245.c9. PMID 17012527